CLINICAL TRIAL: NCT05485051
Title: Impact of Chlorhexidine Bath on Healthcare-associated Infections Acquisitions in Intensive Care Units - A Cluster Randomized Trial
Brief Title: Daily Chlorexidine Bath for Health Care Associated Infection Prevention
Acronym: CLEAN-IT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Collaborators: Hospital Sírio-Libanês (Unknown); Hospital Israelita Albert Einstein (Other); Hospital Moinhos de Vento (Other); Hospital Alemão Oswaldo Cruz (Other); A Beneficência Portuguesa de São Paulo (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: ip_hcor_cleanit
Record Dates: First submitted 2022-07-28; First posted 2022-08-02 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-05

CONDITIONS: Health Care Associated Infection; Ventilator Associated Pneumonia; Central Line-associated Bloodstream Infection (CLABSI); Catheter-Associated Urinary Tract Infection
MeSH Terms: conditions — Cross Infection; Pneumonia, Ventilator-Associated | interventions — Surface-Active Agents; Soaps

STUDY DESIGN:
Intervention Model Description: The study consists in two intervention (chlorhexidine baths) periods (three months each period) and two control (usual baths) periods (three months each period) for each cluster. The clusters will crossover between intervention and control with one month of washout period between different periods.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chlorhexidine baths (Experimental): All patients in the cluster randomized to the intervention arm will receive baths using a 2% chlorhexidine digluconate solution with surface-active agents during the intervention period. All other infection control and cleaning procedures will be performed according to the current practice in each center.
  Interventions: Other: 2% chlorhexidine digluconate solution with surface-active agents
- Usual baths (Active Comparator): All patients in the cluster randomized to the intervention arm will receive baths using soap and water according to the current practice in each center during the intervention period. All other infection control and cleaning procedures will be performed according to the current practice in each center.
  Interventions: Other: Usual Baths

INTERVENTIONS:
Other: 2% chlorhexidine digluconate solution with surface-active agents — Bathing will be performed at least daily using 2% chlorhexidine digluconate solution with surface-active agents on all applicable bathing surfaces, which consists of the entire body surface of the patient except eyes, inner ear, oral mucosa, and areas of loss of skin continuity (such as burnt areas, pressure injuries, etc.); These areas will be bathed according to each center current practice.
  Other Names: Chlorhexidine baths
  Arms: Chlorhexidine baths
Other: Usual Baths — Bathing will be performed at least daily using soap and water (performed according to the current practice in each center) on all applicable bathing surfaces, which consists of the entire body surface of the patient except eyes, inner ear, oral mucosa, and areas of loss of skin continuity (such as burnt areas, pressure injuries, etc.); These areas will be bathed according to each center current practice.
  Other Names: Soap and water baths
  Arms: Usual baths

SUMMARY:
Cluster randomized controlled trial comparing two bathing strategies in critically ill patients. The intervention group will receive daily bathing with chlorhexidine. The control group will receive usual care.

DETAILED DESCRIPTION:
Healthcare-associated infections (HAI) are common complications in critically ill patients and are associated with increased costs, higher length of stay, and higher morbimortality. Data shows that daily chlorhexidine baths might be associated with lower HAI rates in a broad population of critically ill patients. The purpose of this trial is to evaluate the effect of daily bathing with chlorhexidine compared to usual baths (soap and water) on HAI in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients ≥ 18 years/old admitted to the participants's ICUs

Exclusion Criteria:

* History of chlorhexidine allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15730 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Composite of healthcare-associated infections (HAI) | Within each cluster duration (90 days)
  Composite outcome of the following HAI:
  Ventilator associated pneumonia (VAP) Central line-associated blood stream infections (CLABSI) Catheter-associated urinary tract infection (CAUTI)

SECONDARY OUTCOMES:
Rates of multi-drug-resistant pathogens | Within each cluster duration (90 days)
  Rates of positive clinical microbiological cultures (colonization and infection) by multi-drug-resistant (MDR) pathogens.
Ventilator associated pneumonia (VAP) | Within each cluster duration (90 days)
  Rates of Ventilator associated pneumonia (VAP)
Central line-associated blood stream infections (CLABSI) | Within each cluster duration (90 days)
  Rates of Central line-associated blood stream infections (CLABSI)
Catheter-associated urinary tract infection (CAUTI) | Within each cluster duration (90 days)
  Rates of Catheter-associated urinary tract infection (CAUTI)
Hospital length of stay | Until hospital discharge, maximum 90 days
  Hospital length of stay
Intensive Care Unit length of stay | Until Intensive Care Unit discharge, maximum 90 days
  Intensive Care Unit length of stay
Antibiotic use | Within each cluster duration (90 days)
  Antibiotic use per unit
In hospital mortality | Maximum 90 days after randomization
  In hospital mortality
Intensive Care Unit mortality | Maximum 90 days after randomization
  Intensive Care Unit mortality

CONTACTS AND LOCATIONS:
Overall Officials: Bruno M Tomazini, M.D, Principal Investigator — btomazini@hcor.com.br; Alexandre B Cavalcanti, M.D, Study Director — HCor Research Institute Director
Locations (16):
- Brazil (16):
  - Hospital Maternidade São José - UNESC - Fundação Social Rural de Colatina, Colatina, Espírito Santo
  - Hospital da Bahia, Salvador, Estado de Bahia
  - Hospital da Cidade, Salvador, Estado de Bahia
  - Hospital Universitário de Brasília, Brasília, Federal District
  - Hospital Municipal de Maringá, Maringá, Paraná
  - Hospital Regional do Baixo Amazonas Dr. Waldemar Penna, Santarém, Pará
  - Hospital das Clínicas da Universidade Federal de Pernambuco, Recife, Pernambuco
  - Hospital Geral de Caxias do Sul, Caxias do Sul, Rio Grande do Sul
  - Hospital Santa Cruz, Santa Cruz do Sul, Rio Grande do Sul
  - Hospital Nereu Ramos, Florianópolis, Santa Catarina
  - Instituto Baía Sul de Ensino e Pesquisa Irineu May Brodbeck, Florianópolis, Santa Catarina
  - Hospital São Lucas, Aracaju, Sergipe
  - Hospital Aviccena, São Paulo, São Paulo
  - Hospital Naval Marcílio Dias, Rio de Janeiro
  - AC Camargo Câncer Center, São Paulo
  - BP-A Beneficiência Portuguesa de São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: 1 year after publication of primary results
Access Criteria: Submission of a statistical analysis plan for the purposed analyses. Compliance with Brazilian. Data privacy law.